CLINICAL TRIAL: NCT05802368
Title: Adolescents With Hemophilic Knee Arthropathy Can Improve Their Gait Characteristics, Functional Ability, and Physical Activity Level Through Kinect-based Virtual Reality: a Randomized Clinical Trial
Brief Title: Hemophilic Knee Arthropathy Virtual Reality
Acronym: hemophilia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maged Basha (Other)
Collaborators: Cairo University (Other); Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Sponsor-Investigator, Maged Basha, Assistant Professor, College of Medical Rehabilitation, Qassim University, Qassim University
Organization: Qassim University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHPT/0021/0023
Record Dates: First submitted 2023-03-27; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Hemophilia; Knee Arthropathy
MeSH Terms: conditions — Hemophilia A | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): a 30-minute VR-based training session utilizing Kinect Xbox after the session of traditional physical therapy.
  Interventions: Other: virtual reality group; Other: exercise group
- control group (Experimental): Traditional physical therapy, 30-minutes physical therapy exercise program each week with 48-hour intervals at least
  Interventions: Other: exercise group

INTERVENTIONS:
Other: virtual reality group — a 30-minute VR-based training session utilizing Kinect Xbox after the session of traditional physical therapy.
  Other Names: Kinect based virtual reality combined with physical exercises
  Arms: study group
Other: exercise group — Traditional physical therapy, 30-minutes physical therapy exercise program each week with 48-hour intervals at least
  Other Names: physical exercises alone

SUMMARY:
This study intended to examine the effect of a physical rehabilitation program incorporating Kinect-based virtual reality on gait characteristics, functional ability, and physical activity level in adolescents with hemophilic knee arthropathy.

DETAILED DESCRIPTION:
The usage of virtual reality in clinical practice as an alternative for conventional procedures has recently sparked the interest of health professionals. Virtual reality is a type of computer technology that provides simulated sensory feedback to allow children to participate in activities and events that are comparable to those they could face in real life. It can be used therapeutically to enhance strength, range of motion, coordination, mental concentration, problem solving, decision making, balance, and gait.

ELIGIBILITY:
Inclusion Criteria:

* moderate hemophilia
* bilateral involvement of the knee joint
* medically stable and received their factor replacement therapy
* free from contracture or congenital anomalies
* didn't have persisting, disabling pain.

Exclusion Criteria:

* recent bleeding episodes
* severe radiological abnormalities such as bone erosions, degeneration, bone ankylosis, or joint subluxation
* engagement in a regular exercise program in the past six months
* the unwillingness to stick to the training schedule

Ages: 10 Years to 14 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-10-16 (Actual); Study Completion 2023-01-23 (Actual)

PRIMARY OUTCOMES:
Gait Analysis | at first week
  Each participant was instructed to walk bare feet with a comfortable, self-selected speed along a 10-meter walkway while the trajectories of reflective markers and forces were respectively recorded through 12 optoelectronic cameras (Vicon Motion Systems Ltd., Oxford, UK) with a 120-Hz sampling rate and two force plates at 1000 Hz.
Gait Analysis | after 12 weeks
  Each participant was instructed to walk bare feet with a comfortable, self-selected speed along a 10-meter walkway while the trajectories of reflective markers and forces were respectively recorded through 12 optoelectronic cameras (Vicon Motion Systems Ltd., Oxford, UK) with a 120-Hz sampling rate and two force plates at 1000 Hz.

SECONDARY OUTCOMES:
Functional ability assessment | at first week
  The 6-minute walk test was used to assess functional abilities.
Functional ability assessment | after 12 weeks
  The 6-minute walk test was used to assess functional abilities.
Physical activity level assessment | at first week
  The Adolescents' Physical Activity Questionnaire (PAQ-A) in Arabic edition was used to measure the physical activity level assessment.
Physical activity level assessment | after 12 weeks
  The Adolescents' Physical Activity Questionnaire (PAQ-A) in Arabic edition was used to measure the physical activity level assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Alshimaa Azab, PhD, Principal Investigator — Prince Sattam Bin Abdulaziz University
Locations (1):
- King Khalid Hospital, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol
Time Frame: 6 months after publication
Access Criteria: relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.

REFERENCES:
- [Background] Hilberg T, Herbsleb M, Gabriel HH, Jeschke D, Schramm W. Proprioception and isometric muscular strength in haemophilic subjects. Haemophilia. 2001 Nov;7(6):582-8. doi: 10.1046/j.1365-2516.2001.00563.x. PMID 11851757
- [Background] Falk B, Portal S, Tiktinsky R, Weinstein Y, Constantini N, Martinowitz U. Anaerobic power and muscle strength in young hemophilia patients. Med Sci Sports Exerc. 2000 Jan;32(1):52-7. doi: 10.1097/00005768-200001000-00009. PMID 10647529
- [Result] Regaieg S, Charfi N, Yaich S, Damak J, Abid M. The Reliability and Concurrent Validity of a Modified Version of the International Physical Activity Questionnaire for Adolescents (IPAQ-A) in Tunisian Overweight and Obese Youths. Med Princ Pract. 2016;25(3):227-32. doi: 10.1159/000442752. Epub 2015 Nov 26. PMID 26613579